CLINICAL TRIAL: NCT06452602
Title: Induction Immunochemotherapy Followed by Concurrent Chemoradiotherapy for Patients With Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma: a Stratified Exploratory Phase 2 Trial.
Brief Title: Induction Immunochemotherapy Followed by Concurrent Chemoradiotherapy in Patients With ESCC.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20240610
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer
Keywords: Induction Immunochemotherapy; Adebrelimab; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction Immunochemotherapy (Experimental)
  Interventions: Drug: Induction immunochemotherapy followed by Adebrelimab plus concurrent chemoradiotherapy; Drug: Induction immunochemotherapy followed by concurrent chemoradiotherapy

INTERVENTIONS:
Drug: Induction immunochemotherapy followed by Adebrelimab plus concurrent chemoradiotherapy — Induction immunochemotherapy:
  Nab-paclitaxel：220mg/m2，IV，d1，d22; Carboplatin：AUC=5，IV，d1，d22; Adebrelimab：1200mg, IV，d1, d22.
  Evaluation of the Curative Effect：CR+PR
  Adebrelimab plus concurrent chemoradiotherapy:
  Adebrelimab：1200mg, IV，q3w, until PD; Nab-paclitaxel：175mg/m2，IV，d1，d22; Carboplatin：AUC=5，IV，d1，d22; Radiotherapy：50.4Gy/1.8Gy/28f.
  Other Names: Adebrelimab plus concurrent chemoradiotherapy; CR+PR group
Drug: Induction immunochemotherapy followed by concurrent chemoradiotherapy — Induction immunochemotherapy:
  Nab-paclitaxel：220mg/m2，IV，d1，d22; Carboplatin：AUC=5，IV，d1，d22; Adebrelimab：1200mg, IV，d1, d22.
  Evaluation of the Curative Effect：SD+PD
  Concurrent chemoradiotherapy:
  Oxaliplatin：85 mg/m2，IV，d1，d15，d29; Leucovorin：400mg/m2，IV，d1，d15，d29; 5-FU：400mg/m2，IV，d1，d15，d29; 5-FU：1600mg/m2，CIV48h，d1，d15，d29; Radiotherapy：PTV/PGTV:50.4Gy/59.92Gy/28f.
  Other Names: Concurrent chemoradiotherapy; SD+PD group

SUMMARY:
This trial is conducted in patients with unresectable locally advanced esophageal squamous cell carcinoma. The investigators plan to enroll 60 patients with unresectable locally advanced esophageal cancer in Tianjin cancer hospital.

After 2 cycles of induction immunochemotherapy, 60 patients with ESCC will be divided into 2 groups (CR+PR group and SD+PD group) according to the efficacy of induction therapy. Patients in the CR+PR group will be treated with the same immunochemotherapy regimen plus concurrent radiotherapy (50.4Gy/1.8Gy/28f) . And immunotherapy will maintain for a maximum of 1 year. Patients in the SD+PD group will be treated with concurrent chemoradiotherapy (Radiotherapy: PTV/PGTV:50.4Gy/59.92Gy/28f and another chemotherapy regimen). Immunotherapy will not used during chemoradiotherapy because of immunotherapy resistance.

The trial can effectively stratify patients by induction immunochemotherapy, and a more appropriate treatment regimen for patients has the potential to further improve PFS and prolong OS in all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate, cooperated with follow-up visits;
2. Aged 18 years or older, both male and female;
3. Histologically confirmed cT1N2-3M0 or cT2-4bN0-3M0 or cT1-4bN0-3M1( supraclavicular lymph node metastasis) locally advanced ESCC (8th AJCC );
4. Clinically staged as II-IVb inoperable locally advanced ESCC(including non-resectable, or with contraindications to or refusal of surgery);
5. ECOG performance status 0 or 1;
6. Presence of measurable and/or non-measurable lesions as defined by RECIST 1.1;
7. Haven't received any previous systemic anti-tumor therapy (including but not limited to systemic chemotherapy, radiotherapy, molecularly targeted drug therapy, immunotherapy, biologic therapy, topical therapy and other investigational therapeutic agents);
8. Provide fresh or archived tumour tissue samples within 6 months (fresh samples preferred) for biomarker analysis (e.g.PD-L1). Sample types are formalin-fixed, paraffin-embedded [FFPE] tumour tissue blocks or at least 5 unstained, 3-5 μm thick FFPE tumour tissue sections;
9. Expected survival ≥ 3 months;
10. Adequate hematologic function, defined as ANC ≥1500/μl, platelet count ≥100,000/μl and hemoglobin count ≥9.0 g/dl or ≥5.6 mmol/l;
11. Adequate renal function, defined as creatinine ≤1.5× ULN or measured or calculated creatinine clearance ≥60 mL/min for those with creatinine levels >1.5× ULN (Calculated from the Cockcroft-Gault formula);
12. Adequate hepatic function, defined as total bilirubin ≤1.5× ULN and ALT/AST/AKP levels ≤2.5× ULN and albumin ≥2.8 g/dl;
13. Adequate coagulation function, defined as INR ≤1.5× ULN and APTT≤1.5× ULN unless the patient is receiving anticoagulant therapy as long as INR is within the therapeutic range;
14. Women of childbearing potential with a negative urine pregnancy test within 3 days before the first administration of the investigational drugs.
15. Documented informed consent.

Exclusion Criteria:

1. Surgery for esophageal cancer;
2. Esophageal fistulae due to infiltration of the primary tumour;
3. Risk of gastrointestinal bleeding, oesophageal fistula or oesophageal perforation
4. Poor nutritional status, weight loss of ≥10% in the previous 2 months, with no significant improvement after nutritional intervention;
5. Major surgery or severe trauma within 4 weeks prior to first use of study drug;
6. Uncontrollable pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
7. Received or receiving any of the following treatments in the past:

   1. Anti-PD-1 or anti-PD-L1 antibody therapy, chemotherapy, radiotherapy or targeted therapy;
   2. Participation in a study of an investigational agent or device within 4 weeks before the first dose of study treatment;
   3. Systemic treatment with corticosteroids (>10 mg prednisone equivalent dose per day) or other immunosuppressive agents is required for 2 weeks before the first dose of study treatment(except for the use of corticosteroids for local inflammation of the oesophagus and for the prevention of allergy and nausea and vomiting). Other special circumstances need to be communicated to the sponsor.Inhaled or topical steroids and adrenocorticotropic hormone replacement at doses >10mg/day prednisone efficacy dose are permitted if the patient does not have active autoimmune disease;
   4. Received an anti-tumour vaccine or received a live vaccine within 4 weeks before the first dose of study treatment;
8. Any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonitis, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism);Except for patients with vitiligo or those who had asthma or allergies in childhood but did not need any intervention as adults; patients with autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone and type I diabetes mellitus treated with stable doses of insulin may be included;
9. Diagnosis of immunodeficiency, including positive HIV test,other acquired/congenital immunodeficiency diseases, organ transplantation and allogeneic bone marrow transplantation;
10. Diagnosis of uncontrolled cardiac clinical symptoms or disease such as a.NYHA II or above heart failure b.unstable angina c.myocardial infarction within 1 year d.clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
11. Severe infections (CTCAE > Grade 2), such as severe pneumonia requiring hospitalisation, bacteraemia, infectious co-morbidities, etc., within 4 weeks before the first use of study treatment; Baseline chest imaging suggestive of active lung inflammation, signs and symptoms of infection requiring oral or intravenous antibiotic treatment within 2 weeks before the first use of study treatment, except for prophylactic antibiotic use;
12. History of interstitial lung disease or non-infectious pneumonia, or pulmonary insufficiency ≥ grade 3 as confirmed by pulmonary function tests;
13. Active tuberculosis infection detected by history or CT examination, or history of active tuberculosis infection within 1 year before enrollment or more than 1 year previously without regular treatment;
14. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower limit of detection);
15. Presence of abnormal sodium, potassium, and calcium laboratory test values greater than Grade 1 within 2 weeks prior to randomisation that do not improve with treatment;
16. Known hypersensitivity to large protein preparations, or to any of the components of nab-paclitaxel or carboplatin or to any of the components used within their preparations;
17. Pregnant or lactating patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-06 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 2 years
  progression-free survival

SECONDARY OUTCOMES:
OS | up to 2 years
  overall survival
ORR | up to 2 years
  overall response rate
DoR | up to 2 years
  Duration of Response
AE | up to 3 years
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wencheng zhang, M.D., Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China